CLINICAL TRIAL: NCT03920007
Title: A Phase 1/2 Dose Escalation Study of Subretinally Injected ATSN-101 Administered in Patients With Leber Congenital Amaurosis Caused by Biallelic Mutations in GUCY2D
Brief Title: Study of Subretinally Injected ATSN-101 Administered in Patients With Leber Congenital Amaurosis Caused by Biallelic Mutations in GUCY2D
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Atsena Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATSN-101-1; U1111-1200-1308 (Other: UTN)
Record Dates: First submitted 2019-04-10; First posted 2019-04-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Leber Congenital Amaurosis; LCA; LCA1
Keywords: GUCY2D
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinal cone dystrophy 2 | interventions — Prednisone; Prednisolone; Trimethoprim; Polymyxin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ATSN-101 (Experimental): ATSN-101 single dose according to an ascending dose design (dose escalation phase) or ATSN-101 single dose (dose expansion phase)
  Interventions: Drug: ATSN-101; Drug: ATSN-101 Diluent Solution; Drug: Prednisone; Drug: Triamcinalone Acetonide; Drug: 1% Prednisolone; Drug: Trimethoprim/polymyxin B

INTERVENTIONS:
Drug: ATSN-101 — Pharmaceutical form:Solution for intraocular administration Route of administration: Subretinal injection
Drug: ATSN-101 Diluent Solution — Pharmaceutical form:Solution for parenteral use Route of administration: Subretinal injection
Drug: Prednisone — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Triamcinalone Acetonide — Pharmaceutical form:Suspension Route of administration: Peri-ocular injection
Drug: 1% Prednisolone — Pharmaceutical form:Suspension Route of administration: Drops
Drug: Trimethoprim/polymyxin B — Pharmaceutical form:Solution Route of administration: Topical

SUMMARY:
Primary Objective:

To evaluate the safety and tolerability of ascending doses of ATSN-101 administered as a unilateral subretinal injection in patients with Leber Congenital Amaurosis (LCA) caused by autosomal recessive guanylate cyclase 2D (GUCY2D) mutations (GUCY2D-LCA).

Secondary Objective:

To evaluate the efficacy of ascending doses of ATSN-101 administered as a unilateral subretinal injection in patients with GUCY2D-LCA.

DETAILED DESCRIPTION:
Study duration per participant is approximately 112 weeks including: an approximately 56-day screening/baseline period, an approximately 52-week study observation period including 1 treatment day, and an approximately 52-week safety follow-up period. The end of study visit will be approximately 260 weeks after the Investigational Medicinal Product (IMP) administration.

After completion of the main study (ATSN-101-1), participants may have the option to enroll in a separate long-term follow-up study, in which case they would no longer continue in ATSN-101-1 and their end of study visit would be conducted at Week 52.

The study is separated into 2 parts including a dose escalation phase (Part A) and a dose expansion phase (Part B). In Part B participants will be treated at the maximum tolerated dose (MTD) or maximum administered dose (MAD) determined from Part A.

ELIGIBILITY:
Inclusion criteria :

* Male or female participant with clinical diagnosis of Leber congenital amaurosis caused by biallelic mutations in the GUCY2D (retinal guanylate cyclase) gene with all of the following: a) Documented mutations in both alleles of the GUCY2D gene per testing in a CLIA-approved laboratory, b) For Cohort 1-3, best corrected visual acuity (BCVA) of 20/200 or worse in the eye to be injected; subsequent cohorts may include BCVA of 20/80 or worse in the eye to be injected, c) Photoreceptor (outer nuclear) layer structure identifiable on an optical coherence tomography (OCT) scan across the central retina.
* Age ≥18 years for Cohorts 1 through 4, and age ≥ 6 years and <18 years for Cohort 5.
* Male and female participants must follow the contraception requirements of the trial.
* Participants must agree to not donate blood, organs, tissues, cells or sperm for at least three months following ATSN-101 administration.

Exclusion criteria:

* Complicating systemic diseases (such as medical conditions causing immunosuppression) that would preclude the gene transfer, ocular surgery or planned study procedures.
* History of human immunodeficiency virus (HIV) infection.
* Pre-existing eye conditions in the study eye that would preclude the planned surgery or interfere with the assessment and interpretation of study endpoints: for example, glaucoma or optic neuropathy that has resulted in significant visual loss, corneal or lenticular abnormalities or opacities that would preclude view of the fundus or performance of the outcome measures, uveitis, retinopathy and maculopathy that in the opinion of the Investigator are causing significant visual loss.
* Presence of significant ocular abnormalities in the study eye that in the opinion of the Investigator would preclude the planned surgery, effective safety follow-up, or interfere with the interpretation of study endpoints (eg, glaucoma, corneal or significant lens abnormalities or opacities, pre-existing uveitis, intraocular infection, choroidal neovascularization).
* Any contraindication to the planned surgical procedure, such as contraindications to the use of anaesthesia or allergy to medications planned in the peri-operative period.
* Known allergy or hypersensitivity to any component of the investigational medicinal product (IMP), diagnostic agents used during the study or medications planned for use in the peri-operative period, particularly corticosteroids.
* Women who are pregnant (defined as positive beta-Human Chorionic Gonadotropin (HCG) blood or urine test), lactating or breastfeeding.
* Any ocular procedure, either planned or performed within 6 months of Day 1, which would interfere with the planned surgery or the interpretation of study endpoints in the opinion of the Principal Investigator (PI).
* Laboratory test abnormalities or abnormalities in electrocardiogram that in the opinion of the PI would make the participant unsuitable for participation in the study.
* Significant intercurrent illness or infection during the 28 days prior to enrollment.
* Current substance use disorder.
* Use of any investigational agent administered within 5 times the elimination half-life of that investigational agent prior to ATSN-101 administration.
* Enrollment in any other clinical treatment study, for any condition, including those relating to GUCY2D-LCA, throughout the duration of the ATSN-101 study participation.
* Use of anticoagulation therapy within two weeks prior to surgery.
* Use of immunosuppressive medications.
* Current, planned during the course of this trial, or past (within 5 times the elimination half-life of that therapy prior to ATSN-101 administration) use of anti-viral therapy that would inactivate the investigational agent.
* Received gene therapy within the last 15 years.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) from baseline up to the end of the observation period | From baseline to week 52
  Number of participants with AEs will be summarized in each cohort and overall
Number of participants with AEs from baseline up to the end of the safety follow-up period | From baseline to week 260
  Number of participants with AEs will be summarized in each cohort and overall

SECONDARY OUTCOMES:
Change in best -corrected visual acuity (BCVA) | Baseline to week 52 and Baseline to week 260
  Change in BCVA from baseline in the treated and untreated eye (control)
Change in sensitivity | Baseline to week 52 and Baseline to week 260
  Change in sensitivity from baseline in the treated eye and untreated eye (control) as measured by the full-field stimulus testing

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Casey Eye Institute - Oregon Health & Science University, Portland, Oregon
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.clinicalstudydatarequest.com/